CLINICAL TRIAL: NCT01327248
Title: Clinical Status and Bronchial Inflammation in Patients With Bronchiolitis Obliterans
Acronym: Frabo
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Rosewich, Martin Rosewich, MD, Johann Wolfgang Goethe University Hospital
Other Study IDs: FRA-BO
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Bronchiolitis Obliterans
Keywords: Bronchiolitis obliterans; HRCT; Sputum; Blood; Inflammation; adaptive immune system; innate immune system
MeSH Terms: conditions — Bronchiolitis Obliterans; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, and Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- affected patients: 20 Patients suffering from bronchiolitis obliterans
- non-affected patients: 20 matched controls not suffering from bronchiolitis obliterans

SUMMARY:
The aim of this case-control study is the characterization of the bronchial and systemic inflammation of children and young adults with bronchiolitis obliterans.

On the first visit subjects are asked to perform a lung function test (spirometry, body plethysmography with helium). Further levels of eNO and eCO are determined. A blood sample is drawn to describe the inflammatory status. Bronchial inflammation will be measured in induced sputum. At the second visit, a non-specific bronchial provocation testing (PD20 FEV1 methacholine) is performed.

DETAILED DESCRIPTION:
Objectives:

The aim of this study is the characterization of patients with bronchiolitis obliterans in terms of lung function, bronchial hyperreactivity and the degree of the systemic and bronchial inflammation.

Sputum and serum samples are analyzed by quantitative real-time polymerase chain reaction (PCR) (qRT-PCR) and by cytometric bead assay (CBA). Components of the innate immune system (mannose-binding protein, TLR recognition proteins and surfactant proteins) are genetically determined from sputum or blood respectively. In the conduct of this study the investigators will retrospectively and systematically evaluate the available high-resolution computed tomography (HRCT) studies of affected patients

Methods and Work Programme:

This study consists of two study visits (V1 and V2)

V1:

* Measurement of nitric oxide in expired air (eNO)
* Measurement of carbon monoxide in the exhaled air (eCO)
* Lung function testing with spirometry and body plethysmography
* Blood test: blood count, CRP, RAST, serum inflammatory mediators, genetic markers of the non-specific pulmonary defense system
* Induced sputum for inflammatory mediators and microbiological investigations

V2:

• Unspecific bronchial provocation test with methacholine (PD20 FEV1 methacholine)

Study population:

Children and young people (6 - 25 years of age). Both the patients and the healthy subjects are recruited from the outpatient clinic of Pediatric Allergy and Pulmonology.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* between 6 and 25 years of age
* Known bronchiolitis obliterans / no bronchiolitis obliterans(depending on the study group)
* Ability to perform lung function tests and inhalation

Exclusion Criteria:

* <6 and > 25 years of age on the day of written informed consent
* Acute illness with systemic or bronchial inflammation
* every chronic condition or infection (eg HIV, tuberculosis, malignancy)
* pregnancy
* known alcohol and/ or drug abuse
* Inability to understand the extent and scope of the study
* Participation in another study

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study is carried out in children and young adults (6 to 25 years). Both the patients (20) and the healthy subjects (20) are recruited from the outpatient clinic of the departement of Pediatric Allergy and Pulmonology, University Clinic, JW Goethe University, Frankfurt/M, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rosewich, MD, Principal Investigator — Goethe University
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Kurland G, Michelson P. Bronchiolitis obliterans in children. Pediatr Pulmonol. 2005 Mar;39(3):193-208. doi: 10.1002/ppul.20145. PMID 15635614
- [Background] Pichler M, Herrmann G, Schmidt H, Ahrens P, Zielen S. Persistent adenoviral infection and chronic obstructive bronchitis in children: is there a link? Pediatr Pulmonol. 2001 Nov;32(5):367-71. doi: 10.1002/ppul.1145. PMID 11596161
- [Background] Pichler MN, Reichenbach J, Schmidt H, Herrmann G, Zielen S. Severe adenovirus bronchiolitis in children. Acta Paediatr. 2000 Nov;89(11):1387-9. doi: 10.1080/080352500300002633. PMID 11106056
- [Background] Gerhardt SG, McDyer JF, Girgis RE, Conte JV, Yang SC, Orens JB. Maintenance azithromycin therapy for bronchiolitis obliterans syndrome: results of a pilot study. Am J Respir Crit Care Med. 2003 Jul 1;168(1):121-5. doi: 10.1164/rccm.200212-1424BC. Epub 2003 Apr 2. PMID 12672648